CLINICAL TRIAL: NCT05767723
Title: Platelet Function Evaluation in Patients With Acute Coronary Syndromes on Potent P2Y12 Inhibitor Monotherapy Versus Dual Antiplatelet Therapy With Aspirin and a Potent P2Y12 Inhibitor
Brief Title: Platelet Sub-study of the Neomindset Trial
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Platelet
Record Dates: First submitted 2023-02-15; First posted 2023-03-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; antithrombotic therapy; dual antiplatelet therapy; monotherapy
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Aspirin; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetylsalicylic acid + ticagrelor OR Acetylsalicylic acid + prasugrel (Active Comparator): Subjects randomized to Dual Antiplatelet Therapy Control Group will be treated with a regimen of acetylsalicylic acid combined with ticagrelor or prasugrel for 12 months.
  Acetylsalicylic acid (100 mg/day) + ticagrelor (90 mg twice daily) Or Acetylsalicylic acid (100 mg/day) + prasugrel (10 mg once daily)
  Interventions: Drug: Dual antiplatelet therapy: Acetylsalicylic acid + ticagrelor OR Acetylsalicylic acid + prasugrel
- Ticagrelor alone or prasugrel alone (Experimental): All subjects randomized to Monotherapy Group will have acetylsalicylic acid discontinued immediately after randomization.
  Subjects randomized to Monotherapy Group will be treated with ticagrelor (90 mg twice daily) or prasugrel alone (10 mg once daily) for 12 months.
  Ticagrelor alone (90 mg twice daily) Or Prasugrel alone (10 mg once daily)
  Interventions: Drug: Monotherapy: Ticagrelor alone OR Prasugrel alone

INTERVENTIONS:
Drug: Dual antiplatelet therapy: Acetylsalicylic acid + ticagrelor OR Acetylsalicylic acid + prasugrel — Acetylsalicylic acid (100 mg/day) + ticagrelor (90 mg twice daily) Or Acetylsalicylic acid (100 mg/day) + prasugrel (10 mg once daily)
  Other Names: Dual Antiplatelet Therapy
  Arms: Acetylsalicylic acid + ticagrelor OR Acetylsalicylic acid + prasugrel
Drug: Monotherapy: Ticagrelor alone OR Prasugrel alone — Ticagrelor alone (90 mg twice daily) OR Prasugrel alone (10 mg once daily)
  Other Names: Monotherapy
  Arms: Ticagrelor alone or prasugrel alone

SUMMARY:
The general purpose of the Neomindset trial is to evaluate the non-inferiority hypothesis for ischemic events and the superiority hypothesis for bleeding events resulting from platelet P2Y12 receptor inhibitors given as monotherapy in comparison with conventional dual antiplatelet therapy in acute coronary syndrome patients treated with percutaneous coronary intervention.

The platelet sub-study will be conducted at the Hospital Israelita Albert Einstein. This sub-study will recruit randomized patients from the Neomindset trial to evaluate platelet function after at least 30 days of study treatment with either P2Y12 inhibitor monotherapy or dual antiplatelet therapy.

DETAILED DESCRIPTION:
The platelet sub-study will be conducted at the Hospital Israelita Albert Einstein. This sub-study will recruit randomized patients from the Neomindset trial to evaluate platelet function after at least 30 days of study treatment with either P2Y12 inhibitor monotherapy or dual antiplatelet therapy.

These patients will undergo blood sampling and measurement of platelet function after being treated with P2Y12 inhibitor monotherapy or dual antiplatelet therapy for at least 30 days.

ELIGIBILITY:
Inclusion criteria:

* Age >=18 years;
* Clinical presentation compatible with acute coronary syndrome with onset < 24 hours before admission;
* Successful percutaneous coronary intervention(s) of all target lesions (culprit and non-culprit) with new-generation drug-eluting stents;
* Length of stay in hospital at randomization < 96 hours;
* Subjects will be informed about the nature of the study and must agree to comply and give an informed consent in writing using a form approved in advance by the local Ethics Committee.

Exclusion Criteria:

* Acute coronary syndrome on index admission treated in a conservative way or by unsuccessful percutaneous intervention or surgically;
* Presence of residual lesions which are likely to require future treatment in the next 12 months;
* Fibrinolytic therapy < 24 hour before randomization;
* Need of oral anticoagulation with warfarin or new anticoagulants;
* Chronic bleeding diathesis;
* Active or recent major bleeding (in-hospital);
* Prior intracranial hemorrhage;
* Ischemic cerebrovascular accident < 30 days;
* Presence of brain arteriovenous malformation;
* Index event of non-atherothrombotic etiology (i.e., stent thrombosis, coronary embolism, spontaneous coronary artery dissection, myocardial ischemia due to supply/demand imbalance);
* Potential or scheduled cardiac or non-cardiac surgery in the next 12 months;
* Platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3;
* Total white blood count < 3,000 cells/mm3;
* Suspected or documented active liver disease (including laboratory evidence of hepatitis B or C);
* Receiver of heart transplant;
* Known allergies or intolerance of acetylsalicylic acid, clopidogrel, ticlopidine, ticagrelor, prasugrel, heparin or antiproliferative agents from the limus-family of drugs;
* Subject with life expectation lower than 1 year;
* Any significant medical condition that, in the investigator's opinion, could interfere with the ideal participation of the subject in the study;
* Participation in other study in the past 12 months, unless a direct benefit to the subject can be expected.
* Impossibility of being treated with dual antiplatelet therapy for 12 months, based on investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Platelet function using PFA-100 | 30 days of treatment
  Platelet function using PFA-100

SECONDARY OUTCOMES:
Platelet function using CHRONO-LOG | 30 days of treatment
  Platelet function using CHRONO-LOG
Platelet function using Rotem-platelet | 30 days of treatment
  Platelet function using Rotem-platelet
Coagulation test using thromboelastogram | 30 days of treatment
  Coagulation test using thromboelastogram

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A Lemos, MD, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Baber U, Zafar MU, Dangas G, Escolar G, Angiolillo DJ, Sharma SK, Kini AS, Sartori S, Joyce L, Vogel B, Farhan S, Gurbel P, Gibson CM, Fuster V, Mehran R, Badimon JJ. Ticagrelor With or Without Aspirin After PCI: The TWILIGHT Platelet Substudy. J Am Coll Cardiol. 2020 Feb 18;75(6):578-586. doi: 10.1016/j.jacc.2019.11.056. PMID 32057371
- [Background] Johnson TW, Baos S, Collett L, Hutchinson JL, Nkau M, Molina M, Aungraheeta R, Reilly-Stitt C, Bowles R, Reeves BC, Rogers CA, Mundell SJ, Baumbach A, Mumford AD. Pharmacodynamic Comparison of Ticagrelor Monotherapy Versus Ticagrelor and Aspirin in Patients After Percutaneous Coronary Intervention: The TEMPLATE (Ticagrelor Monotherapy and Platelet Reactivity) Randomized Controlled Trial. J Am Heart Assoc. 2020 Dec 15;9(24):e016495. doi: 10.1161/JAHA.120.016495. Epub 2020 Dec 11. PMID 33305660